CLINICAL TRIAL: NCT00000879
Title: A Phase I/II Study to Evaluate the Safety and Immunogenicity of ALVAC HIV Vaccines Alone and With AIDSVAX B/B in Children Born to HIV-Infected Mothers
Brief Title: A Study of the Effects of Giving Two Anti-HIV Vaccines to Babies of HIV-Positive Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: ACTG 326; PACTG 326; 10601 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Pregnancy; Pregnancy Complications, Infectious; AIDS Vaccines; Disease Transmission, Vertical; Avipoxvirus; HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1
Biological: ALVAC-HIV MN120TMG (vCP205)

SUMMARY:
The purpose of this study is to see if giving the ALVAC vCP1452 anti-HIV vaccine alone or with another vaccine called AIDSVAX B/B to babies of HIV-positive mothers is safe. The study will also look at how these vaccines affect a baby's immune system. Most HIV-positive children get HIV from their mothers during pregnancy or birth. Treatment with anti-HIV drugs can reduce the baby's risk of getting HIV. Vaccines also may help prevent HIV infection. This study will look at whether the ALVAC vCP1452 vaccine and the AIDSVAX B/B vaccine can help the body fight off HIV infection. There is no chance of getting HIV infection from the vaccines. (This study has been changed. In earlier versions, ALVAC vCP205 and AIDSVAX B/E were going to be used.)

DETAILED DESCRIPTION:
Transmission of HIV from an untreated infected mother to her offspring is thought to occur to some infants perinatally and others at parturition. It is possible that administration of an immunogenic vaccine can reduce the vertical transmission of HIV-1 or moderate its course in infected infants. Successful early sensitization to HIV epitopes might succeed in preventing HIV infection. Alternately, the enhancement of HIV-specific immune function might also succeed in modifying HIV replication and affecting disease progression.

Sixty infants are treated in this randomized, double-blind study; 45 infants receive recombinant Canarypox virus, ALVAC-HIV vCP205, and 15 receive placebo. Mothers serve as proxy for their infants. All infants receive a minimum of four immunizations, at Weeks 0 (within 72 hours of birth), 4, 8, and 12. Initially, 24 patients are randomized to receive one of two doses of vCP205 or a saline placebo. When a suitable subunit vaccine is available, the protocol will be amended and 36 additional infants will be randomized to receive vCP205 alone or with a subunit vaccine at Weeks 4 and 8 (or vaccine placebo with or without subunit placebo). [AS PER AMENDMENT 11/5/97: 18 infants receive ALVAC-HIV vCP205 at one of two doses and 6 receive placebo.] [AS PER AMENDMENT 9/9/99: Cohort 1 received vCP205. Cohort 2 received a higher dose of vCP205. Cohort A received vCP205 placebo (saline). Cohorts 1, 2, and A were double-blinded and closed to accrual in March 1999. As of September 1999, infants are randomized to one of four new cohorts. Cohort 3 receives vCP1452 at Weeks 0, 4, 8, and 12. Cohort 4 receives vCP1452 at Weeks 0 and 4, then receives vCP1452 plus AIDSVAX B/E gp120 at Weeks 8 and 12. Cohort B receives vCP1452 placebo at Weeks 0, 4, 8, and 12. Cohort C receives vCP1452 placebo at Weeks 0 and 4, then receives vCP1452 placebo plus AIDSVAX B/E placebo at Weeks 8 and 12. All infants are followed every 2 weeks for the first 14 weeks of life, and then every 6 months until age 2. Cord blood is used to establish autologous B cell lines, and CTL assays are performed to characterize the immune response to HIV. In addition, CD4 count, viral load, and mucosal antibody responses are measured. Immunized infants who are not infected with HIV serve as controls for the immunogenicity of the vaccines in the infected infants.] [AS PER AMENDMENT 1/24/00: AIDSVAX B/E has been replaced with AIDSVAX B/B.]

ELIGIBILITY:
Inclusion Criteria

The infant may be eligible if the mother:

* Is HIV-positive.
* Is willing to follow the study guidelines.
* Had her baby at Week 37 of pregnancy or later.

Exclusion Criteria

The infant will not be eligible if the mother:

* Has hepatitis B.
* Is breast-feeding her baby.
* Used certain medications during pregnancy.

The infant will not be eligible if he/she:

* Is more than 3 days old at study entry.
* Has a serious infection or life-threatening illness.

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48
Dates: Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lambert, Study Chair; Daniel Johnson, Study Chair; Stuart Starr, Study Chair
Locations (17):
- United States (17):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Children's Hosp. of Orange County, Orange, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane Univ. Health Science Ctr., Tulane Univ. Hosp. & Clinic, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Univ. of Pennsylvania Health System, Hosp. of the Univ. of Pennsylvania, Philadelphia, Pennsylvania
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Seattle Children's Hospital CRS, Seattle, Washington

REFERENCES:
- [Background] Johnson D, McFarland E, Muresan P, Fenton T, Lambert J, McNamara J, Hawkins E, Bouquin P, Read J, Estep S, Gunurathan S, Gurwith M, PACTG 326 Protocol Team. PACTG 326: A Phase I/II Study to Evaluate the Safety and Immunogenicity of Alvac HIV Vaccines Alone and with AIDSVax B/B in Children Born to HIV-infected Mothers: Preliminary Results. 10th Conference on Retroviruses and Oppurtunistic Infections. Feb 2003. Abstract 404.
- [Result] Lambert JS. HIV vaccines in infants and children. Paediatr Drugs. 2005;7(5):267-76. doi: 10.2165/00148581-200507050-00001. PMID 16220994